CLINICAL TRIAL: NCT06628726
Title: Role of Liver Biopsy As a Diagnostic Tool for Neonatal Jaundice Causes
Brief Title: Liver Biopsy in Diagnosis Neonatal Jaundice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourhan Hassan Fouad Hassan, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: biopsy role neonatal jaundice
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Neonatal Cholestasis; Neonatal Jaundice
Keywords: liver biopsy in neonatal jaundice; Neonatal Cholestasis; liver biopsy
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neonates (Experimental): Neonates with persistent neonatal jaundice underwent liver biopsy
  Interventions: Diagnostic Test: Liver biopsy

INTERVENTIONS:
Diagnostic Test: Liver biopsy — surgical biopsy from liver
  Other Names: Liver wedge biopsy; Liver core biopsy; Liver incisional biopsy

SUMMARY:
1. Identification and characterization of histopathological features of liver in cases of PNJ.
2. Assessment of key histological features in liver biopsy as diagnostic parameters in differentiating intra-hepatic and extra-hepatic causes of PNJ.
3. Evaluation of role of liver biopsy as a diagnostic tool in conjunction with clinical and laboratory findings.

DETAILED DESCRIPTION:
Neonatal cholestasis (NC) is described as an early-life defect in bile production or flow that causes the liver to retain biliary substances. Persistent Neonatal Jaundice (PNJ) is the presence of variable degrees of jaundice, choluria and hypocholic or acholic stools for more than 10 days during early months of life. The rate of neonatal cholestasis is estimated to be 1 per 2,500 live births worldwide.

In Egypt, about 20.4% of full-term newborns develop jaundice yearly. Extrahepatic cholestasis(EHC) and intrahepatic cholestasis(IHC) are the two main causes of persistent neonatal jaundice. This division is according to the presence or absence of extrahepatic obstruction to bile flow. Biliary atresia(BA) and idiopathic neonatal hepatitis(INH) are the most frequent etiologies for EHC and IHC respectively.

It is critical to identify the underlying cause of PNJ in order to start the right surgical or medicinal treatment. Early surgical referral is necessary in biliary atresia(BA) to increase success rates. In the case of treatable metabolic diseases, a prompt diagnosis justifies prompt, targeted therapy and a better prognosis.

Despite the development of new diagnostic means and advances in imaging techniques, non-invasive biomarkers and genomic studies, a liver biopsy done at the right time is still an important tool to evaluate and diagnose patients with cholestasis, as it will help to decide the etiology, the prognosis and eventually the treatment of the patient.

The evaluation of liver biopsies in infantile cholestasis disorders is crucial as the histologic features of many of these disorders may overlap and vary with age.

ELIGIBILITY:
Inclusion Criteria:

* All cases presented with persistent neonatal jaundice in the first year of life in 5 years interval (2019-2023), received at Surgical Pathology Laboratory at Assiut University Hospitals, Egypt.

Exclusion Criteria:

* Patients older than one year.
* Patients who underwent liver biopsy in the same age group but were not diagnosed as Persistent Neonatal Jaundice.
* Patients with deficient clinical data.

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of the key histopathological features in liver biopsy | baseline
  Identification of the key histopathological features in liver biopsy that aid in differentiation intra-hepatic and extra-hepatic causes of persistent neonatal jaundice (PNJ).

SECONDARY OUTCOMES:
Evaluation of significance of liver biopsy as a diagnostic tool | baseline
  Evaluation of significance of liver biopsy as a diagnostic tool with clinical and laboratory findings in detection of persistent neonatal jaundice (PNJ) causes.

CONTACTS AND LOCATIONS:
Overall Officials: Moemen M Hafez, M.D., Study Director — Faculty of Medicine, Assiut University, Assiut, Egypt; Abeer M Refaiy, M.D., Study Director — Faculty of Medicine, Assiut University, Assiut, Egypt

REFERENCES:
- [Background] Mansour E, Eissa AN, Nofal LM, Kharboush I, Reda AA. Morbidity and mortality of low-birth-weight infants in Egypt. East Mediterr Health J. 2005 Jul;11(4):723-31. PMID 16700389
- [Background] Fawaz R, Baumann U, Ekong U, Fischler B, Hadzic N, Mack CL, McLin VA, Molleston JP, Neimark E, Ng VL, Karpen SJ. Guideline for the Evaluation of Cholestatic Jaundice in Infants: Joint Recommendations of the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition and the European Society for Pediatric Gastroenterology, Hepatology, and Nutrition. J Pediatr Gastroenterol Nutr. 2017 Jan;64(1):154-168. doi: 10.1097/MPG.0000000000001334. PMID 27429428
- [Background] Ali KM, Zalata KR, Barakat T, Elzeiny SM. Pathologic approach to Neonatal cholestasis with a simple scoring system for biliary atresia. Virchows Arch. 2024 Jan;484(1):93-102. doi: 10.1007/s00428-023-03704-5. Epub 2023 Nov 27. PMID 38008855